CLINICAL TRIAL: NCT03910959
Title: Therapeutic Effects of Animal-assisted Therapy for Patients in a Minimally Conscious State: a Randomized, Controlled Cross-over Study
Brief Title: Therapeutic Effects of Animal-assisted Therapy for Patients in a Minimally Conscious State
Acronym: MCS Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Dr. Karin Hediger, Principal Investigator, University of Basel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-00350
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Minimally Conscious State
MeSH Terms: conditions — Persistent Vegetative State | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: The study has a randomized, controlled cross-over design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Animal-assisted therapy (Experimental): Patients receive three weeks of two AAT sessions, each lasting ca 30 minutes.
  Interventions: Other: Animal-assisted therapy
- treatment as usual (Active Comparator): Patients receive three weeks of two control sessions, each lasting ca 30 minutes.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Animal-assisted therapy — Therapy in the presence and with interaction with an animal. Involved animals can be all species that live at REHAB Basel and are part of the AAT program. All animals are trained for the specific service with vulnerable patients.
  Arms: Animal-assisted therapy
Other: Conventional therapy — Parallelled conventional therapy sessions (treatment as usual)
  Arms: treatment as usual

SUMMARY:
The aim of this study is to investigate the effects of animal-assisted occupational therapy on patient's consciousness, measured via the achievement of predefined, patient-specific goals.

30 patients in a minimally conscious state will be included in this trial with randomized, controlled cross-over design. Patients will be randomized and allocated to either study arm 1 or 2 with an allocation ratio 1/1. In study arm 1, patients (N=15) receive three weeks of two AAT sessions per week followed by three weeks of two control sessions (TAU) per week. In study arm 2, patients (N=15) receive three weeks of two control sessions (TAU) per week followed by three weeks of two AAT sessions per week. Each session lasts 30 minutes. Goal attainment and secondary outcomes will be measured before the study start (pre-measurement, t0), at the end of the first 3 weeks therapy (post-measurement I, t1), at the start of the second 3 weeks (pre-measurement II, t2) as well as at the study end (post-measurement II, t3).

DETAILED DESCRIPTION:
Early rehabilitation is crucial for patients in a minimally conscious state (MCS). The reorganization of neuronal structures and the recovery of cognitive processes as well as emotional and physical functions are most important. To reach these goals, animal-assisted therapy (AAT) is part of the therapeutic concept at REHAB Basel. Regarding the results of our previous studies at REHAB Basel, patients with brain-injuries can profit from animal-assisted therapy in terms of socioemotional skills and therapy motivation. Furthermore, patients with severe disorder of consciousness showed more behavioural reactions and arousal during AAT compared to standard therapy sessions. However, there is no research investigating if AAT can help to facilitate reaching rehabilitation goals in patients in a MCS and therefore advance neurorehabilitation. Hence, this study investigates if animal-assisted occupational therapy can facilitate attainment of therapeutic goals.

The main outcome is the amount of achievement of predefined, patient-specific therapeutic goals. This will be measured via the JFK Coma Remission Scale revised (CSR-R), the Basler Vegetative State Assessment (BAVESTA) and on a goal attainment scale in %, filled out by the therapist.

Secondary outcomes are:

1. Behavioural reactions via behavioral video coding
2. Heart rate, Heart rate variability (HR/HRV)
3. Electrodermal activity (EDA) / Galvanic skin response (GSR)

The investigators will include 30 patients fulfilling the following inclusion criteria: Inpatients of REHAB Basel in a minimally conscious state (defined via the CRS-R according to the Aspen criteria); Minimum age of 18 years; Informed consent documented by signature by the patient's legal representative. The presence of any one of the following exclusion criteria will lead to exclusion of the participant: Medical contraindications for contact with animals such as allergy, phobia etc.); Enrollment of the investigator, his/her family members, employees and other dependent persons.

The study has a randomized, controlled cross-over design including 30 patients in a minimally conscious state. Patients will be randomized and allocated to either study arm 1 or 2 with an allocation ratio 1/1. In study arm 1, patients (N=15) receive three weeks of two AAT sessions per week followed by three weeks of two control sessions (TAU) per week. In study arm 2, patients (N=15) receive three weeks of two control sessions (TAU) per week followed by three weeks of two AAT sessions per week. Each session lasts 30 minutes. Before starting the study arm 1 or 2 therapists will define individual therapy goals for each patient.

Measurements will be taken before the study start (pre-measurement, t0), at the end of the first 3 weeks therapy (post-measurement I, t1), at the start of the second 3 weeks (pre-measurement II, t2) as well as at the study end (post-measurement II, t3).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of REHAB Basel in a minimally conscious state
* Minimum age of 18 years
* Informed consent documented by signature by the patient's legal representative

Exclusion Criteria:

* Medical contraindications for contact with animals such as allergy, phobia etc.,
* Enrollment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Amount of goal achievement l: CSR-R | 3 weeks
  The goal achievement will be assessed via the JFK Coma Remission Scale revised (CSR-R), with 6 subscales and a total score ranging from 0 to 23 with higher scores indicating better outcomes.
Amount of goal achievement II: BAVESTA | 3 weeks
  The goal achievement will be assessed via the Basler Vegetative State Assessment. The scale ranges from 0 to 5 with higher scores indicating better outcomes.
Amount of goal achievement III: VAS | 3 weeks
  The goal achievement will also be assessed via a Visual Analogue Scale where a cross can be made on a line (measured in millimeters, ranging from 0 to 25) with higher values indicating better outcome.

SECONDARY OUTCOMES:
Behavioral reactions | 3 weeks
  Behaviour of the patients will be coded in Noldus Observer according to a strict ethogram. State behaviours will be reported in % (relative to the duration of a session) and count behaviours as total number of shown behaviours during a session.
Heart rate | 3 weeks
  Heart rate will be measured in peats per minute using a Polar belt. HR is reported in beat per minutes (bpm).
Heart rate variability | 3 weeks
  Heart rate variability will be measured using a Polar belt. HRV is reported as mean RR intervals. The following HRV parameters will be calculated: time domain: the standard deviation of all normal-to-normal RR intervals (SDNN, ms) and root-mean square differences of successive RR intervals (RMSSD, ms); and frequency domain: relative power of the low frequency (LF) and high frequency (HF) band in normal units
Electrodermal activity (Galvanic Skin Response) | 3 weeks
  Electrodermal activity will be measured using the EMBRACE wristband. The outcome is reported in Microsiemens (sampling rate of 4Hz).

CONTACTS AND LOCATIONS:
Locations (1):
- REHAB Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided